CLINICAL TRIAL: NCT00445653
Title: Molecular Epidemiology of Barrett's Esophagus
Brief Title: Risk Factors for Barrett's Esophagus in Patients With BE, Gastroesophageal Reflux, or Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Christopher Christiani, Pulmonary Associate, Massachusetts General Hospital
Other Study IDs: CDR0000450146; MGH-1999-P-010929/13 (Other: Partners Healthcare IRB)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Precancerous Condition
Keywords: Barrett esophagus
MeSH Terms: conditions — Precancerous Conditions; Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples only were collected
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: A study that evaluates DNA changes and other disease-related health information in patients with Barrett's esophagus, gastroesophageal reflux, or gastrointestinal bleeding may help doctors learn more about the risk factors for Barrett's esophagus.

PURPOSE: This clinical trial is looking at DNA changes and other disease-related health information as risk factors for Barrett's esophagus in patients with Barrett's esophagus, gastroesophageal reflux, or gastrointestinal bleeding.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the role of several genetically determined factors that, in combination with CagA status, cigarette smoking, alcohol, and diet to varying degrees, result in an increased risk for Barrett's esophagus.

OUTLINE: This is a controlled study.

Patients complete questionnaires about demographics, medical history, smoking and alcohol history, current medications, frequency and chronicity of gastroesophageal reflux symptoms, and diet history.

Blood and tissue are collected and analyzed by DNA-based assays and enzyme-linked immunosorbent assay for CagA status and polymorphisms in detoxifying enzyme systems, other xenobiotic metabolism pathways (e.g., CYP1A1, CYP2E1, CYP3A4, CYP3A5, NQO, NAT-2), inflammatory gene pathways (e.g., IGF, IGFBF3), and in DNA repair genes or p53 pathways (e.g., XRCC1, p53 gene).

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing elective esophagogastroduodenoscopy for any of the following reasons:

  * Surveillance of Barrett's esophagus
  * Evaluation of severe or refractory gastroesophageal reflux disease or chest pain thought to be due to reflux
  * Gastrointestinal bleeding

PATIENT CHARACTERISTICS:

* Not pregnant

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming in for EGD
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2005-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Polymorphisms in detoxifying enzyme systems such as glutathione S-transferases (e.g., mu, theta, pi) | 2000-2013
Polymorphisms in other xenobiotic metabolism pathways (e.g., CYP1A1, CYP2E1, CYP3A4/5, NQO1, mEH, NAT-2) | 2000-2013
Polymorphisms in inflammatory gene pathways (e.g., MPO, MnSOD, IGF, IGFBF3, Il1-beta) | 2000-2013
Polymorphisms in DNA repair genes or the p53 pathways (e.g., ERCC2, XRCC1, p53, p73, CCND1, p21) | 2000-2013

CONTACTS AND LOCATIONS:
Overall Officials: David C. Christiani, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Harvard School of Public Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No